CLINICAL TRIAL: NCT06415825
Title: Preliminary Muscle Contraction in the Rehabilitation and Prevention of Degenerative Pain in the Spine, Hip, Knee, Ankle, Shoulder, Elbow, and Ankle Joints, as Well as After Hip and Knee Arthroplasty
Brief Title: Preliminary Muscle Contraction in the Rehabilitation and Prevention of Degenerative Pain in the Locomotor System
Acronym: PMQRPDP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Sofia (Other)
Responsible Party: Principal Investigator, Assen Aleksiev, Head of Physical Medicine and Rehabilitation Department, Medical University of Sofia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 757/29012024
Record Dates: First submitted 2024-03-29; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Pain, Back; Pain, Neck; Pain, Hip Burning; Pain, Shoulder; Arthropathy of Knee; Arthropathy of Hip; Pain Syndrome
Keywords: degenerative pain; spine; hip; knee; ankle; shoulder; elbow; hip and knee arthroplasty
MeSH Terms: conditions — Back Pain; Neck Pain; Pain; Shoulder Pain; Somatoform Disorders

STUDY DESIGN:
Intervention Model Description: Both groups will receive standard advice. The maneuver group will receive additional advice - preliminary contraction of the muscles in the corresponding kinesiology segment. This advice will be embedded in all motor activities of daily living involving the relevant area.
Who Masked: Participant
Masking Description: Participants will not know which group they will be in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With pre-contr. (Experimental): The patients will receive standard advice and an additional one - preliminary contraction of the muscles in the corresponding kinesiology segment.
  Interventions: Behavioral: Standard advice and Preliminary muscle contraction; Behavioral: Standard advice
- Without pre-contr. (Active Comparator): The patients will receive standard advice.
  Interventions: Behavioral: Standard advice

INTERVENTIONS:
Behavioral: Standard advice and Preliminary muscle contraction — The maneuver groups will receive standard advice and an additional one - preliminary contraction of the muscles in the corresponding kinesiology segment. This advice will be embedded in all motor activities of daily living involving the relevant area.
  Arms: With pre-contr.
Behavioral: Standard advice — Standard advice includes avoiding heavy physical activity, sudden and unexpected loads, repetitive and prolonged overloads, and long periods of hypomobility.

SUMMARY:
RESEARCH OBJECTIVE: To investigate the effect of muscle preliminary contraction in the rehabilitation and prevention of degenerative pain in the spine, hip, knee, ankle, shoulder, elbow, and ankle joints, as well as after hip and knee arthroplasty. HYPOTHESIS: Muscle preliminary contraction has a significant short-term and long-term effect in the rehabilitation and prevention of degenerative pain in the spine, hip, knee, ankle, shoulder, elbow, and ankle joints, as well as after hip and knee arthroplasty. RESEARCH METHODS: At least 216 patients with degenerative pain in the spine, hip, knee, ankle, shoulder, elbow, and ankle joints, as well as after hip and knee arthroplasty, will be studied. They will be randomized into pairwise sub-groups. All will receive standard advice. The maneuver sub¬groups will receive additional advice - preliminary contraction of the muscles in the corresponding kinesiology segment. This advice will be embedded in all motor activities of daily living involving the relevant area. The following follow-up parameters will be used: visual analogue pain scale, manual muscle testing, goniometry, centimeter, and preliminary contraction success rate. Their follow-up will be threefold - at the beginning, after 1, and after 6 months. For statistical processing, multiple analysis of variance (MANOVA), with post hoc Bonferroni multiple tests, and Pearson correlation analysis, with post hoc regression analysis, will be used. CONCLUSION: The positive results will allow the preliminary muscle contraction to be used as a universal tool in the rehabilitation, prevention, and prevention of degenerative pain in the spine, hip, knee, ankle, shoulder, elbow, and ankle joints, as well as after hip and knee arthroplasty (international contribution). This maneuver is very short (seconds), easy (everybody can perform it), does not require the allocation of time, space, and resources (including financial ones), and is instantly incorporated into everyday life.

DETAILED DESCRIPTION:
RESEARCH OBJECTIVE: To investigate the effect of muscle preliminary contraction in the rehabilitation and prevention of degenerative pain in the spine, hip, knee, ankle, shoulder, elbow, and ankle joints, as well as after hip and knee arthroplasty. SCIENTIFIC IDEA: Muscle latency (M1, M2, triggered response, proprioceptive visual/vestibular responses, and M3) leads to chronic damage. During the first 50-200 milliseconds of the movement, there is no internal muscular protective counterforce against external loads on discs, joints, ligaments, insertions, etc. inert structures (including arthroplastic ones), happening thousands of times a day. This leads to repetitive cumulative microtrauma with damage to the "pneumatic hammer" principle, as well as faster wear in arthroplasties. Precontraction of muscles eliminates latency and stabilizes inert (and arthroplastic) structures. WORKING HYPOTHESIS: Muscle preliminary contraction has a significant short-term and long-term effect in the rehabilitation and prevention of degenerative pain in the spine, hip, knee, ankle, shoulder, elbow, and ankle joints, as well as after hip and knee arthroplasty. RESEARCH METHODS: At least 216 patients with degenerative pain in the spine, hip, knee, ankle, shoulder, elbow, and ankle joints, as well as after hip and knee arthroplasty, will be studied. They will be randomized into pairwise sub-groups. All will receive standard advice. The maneuver sub¬groups will receive additional advice - preliminary contraction of the muscles in the corresponding kinesiology segment. This advice will be embedded in all motor activities of daily living involving the relevant area. The following follow-up parameters will be used: visual analogue pain scale, manual muscle testing, goniometry, centimeter, and preliminary contraction success rate. Their follow-up will be threefold - at the beginning, after 1, and after 6 months. For statistical processing, multiple analysis of variance (MANOVA), with post hoc Bonferroni multiple tests, and Pearson correlation analysis, with post hoc regression analysis, will be used. CONCLUSION: The positive results will allow the preliminary muscle contraction to be used as a universal tool in the rehabilitation, prevention, and prevention of degenerative pain in the spine, hip, knee, ankle, shoulder, elbow, and ankle joints, as well as after hip and knee arthroplasty (international contribution). This maneuver is very short (seconds), easy (everybody can perform it), does not require the allocation of time, space, and resources (including financial ones), and is instantly incorporated into everyday life.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years;
* legal capacity;
* patients with recurrent degenerative pain (at least two relapses in the last 12 months), in various joints (vertebral, hip, knee, ankle, shoulder, elbow, and knee), in an exacerbation stage (started up to 2 weeks before recruitment), occurring with periodic exacerbations and remissions (relapse duration of more than 24 hours, preceded and separated by remission of at least 1 month);
* with excitatory (painful) symptoms (but without ablated ones - without paresis, paralysis, and pelvic-reservoir damage);
* as well as after hip and knee arthroplasty.

Exclusion Criteria:

* age under 18,
* incapacity;
* neurological symptoms have disappeared (paresis, paralysis, and pelvic-reservoir disorders),
* macro-injuries (fractures, dislocations, distortions),
* structural anomalies, severe osteoporosis, infectious diseases, febrility, malignant diseases, specific inflammatory and autoimmune diseases (such as rheumatoid arthritis, ankylosing spondylarthritis, etc.), mental diseases, increased tendency to bleed (hemophilia, etc.), as well as cardiovascular vascular, respiratory, liver, kidney and metabolic damage with marked failure.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-05-14 (Estimated); Primary Completion 2025-05-14 (Estimated); Study Completion 2026-05-14 (Estimated)

PRIMARY OUTCOMES:
Visual analogue pain scale | At baseline, at 1 month, and at 6 months.
  To assess the intensity of pain on a visual analog scale, a 10 centimeters segment is drawn on a piece of paper. The patient notes the intensity of pain on this line between the left end of the line (0=no pain) and the right end (10=maximum pain intensity). The result is registered in centimeters - from 0 to 10 centimeters.

SECONDARY OUTCOMES:
Preliminary muscle contraction success rate | At baseline, at 1 month, and at 6 months.
  Success rate refers to how often patients remember to perform preliminary muscle contraction. For example, if this maneuver is skipped every second movement (standing, sitting, bending, standing, lifting, etc.), the success rate is 50%, every third - 77%, every fourth - 85%, and so on.
Manual muscle testing | At baseline, at 1 month, and at 6 months.
  Muscle strength is verified against the examiner's manual resistance and grading on a 0 to 5 scale accordingly: 0 - No movement; 1 - Flicker of movement; 2 - Through full range actively with gravity counterbalanced; 3 - Through full range actively against gravity; 4 -Through full range actively against some resistance; 5 - Through full range actively against strong resistance. For statistical comparability and prognostic value, this scale will be transformed into percentages of the norm: 0=0%; 1=14.29%; 2=35.72%; 3=57.14%; 4=78.57%; 5=100%.
Range of motion | At baseline, at 1 month, and at 6 months.
  Each specific joint has a range of motion that is expressed in degrees measured by goniometer. For statistical comparability and prognostic value, the angular degrees will be transformed into percentages of the norm from 0 to 100%.
Centimeter measurements | At baseline, at 1 month, and at 6 months.
  Centimeter measurements of circumferences of kinetic segments for verification of muscle hypotrophy - in centimeters.
Thomayer's test | At baseline, at 1 month, and at 6 months.
  Thomayer's test is performed from a standing position with maximum flexion of the torso, bending the body forward and down with relaxed arms to the floor. The distance from the tip of the extended fingers to the floor is measured in centimeters. Inability to reach the floor with fingers is considered limited ROM (centimeters with a negative sign), when touching the floor with fingers - normal ROM (0 centimeters), and when touching the floor with palms - hypermobility (centimeters with a positive sign).
Schober's test | At baseline, at 1 month, and at 6 months.
  Schober's test is performed from a standing position. A 15 cm descending segment from the processus spinosus of L1 (in the caudal direction) is measured and the two points are marked. Maximum flexion of the torso is performed by bending the body forward and downward. From the final flexion position, the distance between the two marked points is measured. The increase in the distance between the two points is recorded. The reference values are from 2.5 to 5 cm., i.e. under 2.5 cm. is considered hypomobility, and over 5 cm. - hypermobility.
Ott's test | At baseline, at 1 month, and at 6 months.
  Ott's test is performed from a standing position. A 30 cm descending segment from the processus spinosus of C7 is measured (in the caudal direction) and the two points are marked. Maximum flexion of the torso is performed by bending the body forward and downward. From the final flexion position, the distance between the two marked points is measured. The increase in the distance between the two points is registered. Reference values are from 2.5 to 5 cm., i.e. under 2.5 cm. is considered hypomobility, and over 5 cm. - hypermobility.

CONTACTS AND LOCATIONS:
Overall Officials: Assen R Aleksiev, Principal Investigator — Head Department of Physical Medicne and Rehabilitation, Medical University of Sofia

IPD SHARING:
Plan to Share IPD: Yes
All global statistical data except personal information from the patients.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available from 11.05.2025 to 11.05.2026.
Access Criteria: The data will become available upon request from the principal investigator.

REFERENCES:
- [Background] Aleksiev AR. Ten-year follow-up of strengthening versus flexibility exercises with or without abdominal bracing in recurrent low back pain. Spine (Phila Pa 1976). 2014 Jun 1;39(13):997-1003. doi: 10.1097/BRS.0000000000000338. PMID 24732860
- [Background] Magnusson ML, Aleksiev A, Wilder DG, Pope MH, Spratt K, Lee SH, Goel VK, Weinstein JN. European Spine Society--the AcroMed Prize for Spinal Research 1995. Unexpected load and asymmetric posture as etiologic factors in low back pain. Eur Spine J. 1996;5(1):23-35. doi: 10.1007/BF00307824. PMID 8689414
- [Background] Wilder DG, Aleksiev AR, Magnusson ML, Pope MH, Spratt KF, Goel VK. Muscular response to sudden load. A tool to evaluate fatigue and rehabilitation. Spine (Phila Pa 1976). 1996 Nov 15;21(22):2628-39. doi: 10.1097/00007632-199611150-00013. PMID 9045348